CLINICAL TRIAL: NCT03718143
Title: A Phase 2 Study of WEE1 Inhibition and AZD1775 Alone or Combined With Cytarabine in Patients With Advanced Acute Myeloid Leukemia, Myelodysplastic Syndrome and Myelofibrosis
Brief Title: AZD1775 in Advanced Acute Myeloid Leukemia, Myelodysplastic Syndrome and Myelofibrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Safety concerns
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-01816
Record Dates: First submitted 2018-10-08; First posted 2018-10-24 (Actual); Results first posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Myelofibroses; Acute Myeloid Leukemia; Myelodysplastic Syndromes
MeSH Terms: conditions — Primary Myelofibrosis; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Elderly Newly diagnosed AML (Experimental): Combination AZD1775 with AraC
  Elderly, newly diagnosed AML
  Interventions: Drug: Combination AZD1775 with AraC
- Arm B:Relapsed AML and MDS (Experimental): Combination AZD1775 with AraC
  Relapsed/Refractory AML & HMA failure AML/ MDS
  Interventions: Drug: Combination AZD1775 with AraC
- Arm C: Relapsed AML, MDS and MF (Active Comparator): AZD1775 only
  Relapsed/Refractory AML & HMA failure AML/ MDS and Relapsed/Refractory Primary & Secondary MF
  Interventions: Drug: AZD1775 only

INTERVENTIONS:
Drug: Combination AZD1775 with AraC — AZD1775 days 1-5 & 8-12 AraC days 1-5 & 8-12
  Arms: Arm A: Elderly Newly diagnosed AML; Arm B:Relapsed AML and MDS
Drug: AZD1775 only — AZD1775 days 1-5 & 8-12
  Arms: Arm C: Relapsed AML, MDS and MF

SUMMARY:
A phase II study testing the efficacy of combined AZD1775 with AraC or single agent activity of AZD1775 in three arms: Arm A has subjects age 60 years or older who are newly diagnosed with AML receiving the combination of the drugs; Arm B has subjects who are have relapsed/refractory AML and HMA failure MDS patients being allocated to either the combination Arm B or single agent AZD1775 Arm C.

DETAILED DESCRIPTION:
A phase II study testing the clinical efficacy of combined AZD1775 with AraC or single agent activity of AZD1775 in three patient strata: Elderly(> 60 years) newly diagnosed AML patients (Arm A) will only receive the combination; whereas relapsed/refractory AML patients and HMA failure MDS patients will be allocated to either the combination (Arm B) or single agent AZD1775 (Arm C). The study will have a run in safety cohort of six patients in each of the three arms to determine the safe use of combined AraC /AZD1775 or single agent AZD1775 in the patient populations. This will be followed by an expansion phase of up to 20 and 21 eligible patients in each arm respectively where elderly patients with newly diagnosed AML will receive a combination of AZD1775 and AraC (Arm A) while patients with relapsed or refractory AML or HMA failure MDS will be allocated to receive either AZD1775 with AraC (Arm B) or AZD1775 alone (Arm C). An early toxicity check will be conducted to determine safety and tolerability. If indicated, dose levels will be reduced. The study will continue to enroll the rest of the patients at the tolerated dose.

ELIGIBILITY:
Inclusion:

Inclusion Criteria

* Dose escalation part of trial for combined AraC + AZD1775 (Arm A)
* untreated elderly (>60 years) AML if in the poor-risk cytogenetic group (please reference Appendix V).
* untreated elderly (>60 years) AML if in the intermediate and poor-risk cytogenetic group (please reference Appendix V)
* relapsed or refractory AML (≥ 18 years)
* any MDS (≥ 18 years) having failed or been intolerant to prior hypomethylating agent (HMA) treatment.
* Failure is defined as any disease progression while on HMA, relapse after HMA treatment or no response after 4 cycles of 5-Azacitidine or decitabine
* Patients with isolated 5q-/5q- syndrome must have failed, not tolerated, or progressed on lenalidomide in addition to having failed or been intolerant to HMA treatment.
* advanced progressive MF, defined as intermediate and high risk primary and secondary MF, or any other MF failed or intolerant to JAK2 inhibitor therapy requiring medical therapy
* If appropriate, patients can have failed other prior therapies for their disease (i.e. JAK2 inhibitor, interferon, hydroxyurea or IMIDs). Patients may have failed more than one JAK2 inhibitor and JAK2 inhibitor must not have been the most recent treatment (e.g. other therapies as last therapy prior to study given after failure of previous JAK2 inhibitor).
* Failure/ intolerance of Ruxolitinib
* The following laboratory values obtained 7 days prior to registration.
* Total bilirubin ≤ 1.5 mg/dL (except Gilbert's syndrome or known hemolysis or leukemic infiltration)
* AST (SGOT) and ALT (SGPT) ≤ 2.5 x Upper Limit normal (ULN) or < 5 x ULN if organ involvement
* Alkaline Phosphatase < 5 x ULN - Serum creatinine ≤1.5 x ULN, or measured creatinine clearance (CrCl) ≥45 mL/min as calculated by the Cockcroft-Gault method (confirmation of creatinine clearance is only required when creatinine is >1.5 x institutional ULN) CrCl (glomerular filtration rate [GFR]) = (140-age) x (weight/kg) x Fa (72 x serum creatinine mg/dL) a where F= 0.85 for females and F=1 for males
* ECOG Performance Status (PS) 0, 1 (Appendix I).
* Ability to provide informed written consent and be able to adhere to the study visit schedule and other protocol requirements.
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study).
* Willing to provide blood and bone marrow aspirate samples for correlative research purposes
* Negative serum pregnancy test done ≤7 days prior to registration, for women of childbearing potential only.
* Female patients who are not of child-bearing potential and fertile females of childbearing potential
* Male patients should be willing to abstain or use barrier contraception (i.e., condoms) for the duration of the study drug exposure and for 3 months after study treatment discontinuation.
* Patients who have undergone stem cell transplantation (SCT), autologous or allogeneic, are eligible provided that they are > 60 days from stem cell infusion, have GVHD < grade 1 and are off immunosuppressive agents for > 28 days at time of registration.

Exclusion:

* AML patients who are suitable for and willing to receive intensive chemotherapy
* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Subject has had prescription or non-prescription drugs or other products known to be sensitive CYP3A4 substrates or CYP3A4 substrates
* The preferred azole anti-fungal medication is Fluconazole (alternatively Posaconazole) which can be given during treatment with AZD1775 (section 9.5).
* Pateints may not be on an inhibitor of BCRP as outlined in Appendix VI.
* Not willing to avoid grapefruit, grapefruit juices, grapefruit hybrids, Seville oranges, pummelos, and exotic citrus fruits from 7 days prior to the dose of study medication
* Mean resting corrected QTc interval using the Fridericia formula (QTcF) >450 msec/male and >470 msec/female (as calculated per institutional standards) obtained from 3 electrocardiograms (ECGs) 2-5 minutes apart at study entry, or congenital long QT syndrome
* Herbal preparations/medications

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices). Upon reasonable request.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Elderly Newly Diagnosed AML: Combination AZD1775 with AraC
  Elderly, newly diagnosed AML
  Combination AZD1775 with AraC: AZD1775 days 1-5 & 8-12 AraC days 1-5 & 8-12
- Arm B:Relapsed AML and MDS: Combination AZD1775 with AraC
  Relapsed/Refractory AML & HMA failure AML/ MDS
  Combination AZD1775 with AraC: AZD1775 days 1-5 & 8-12 AraC days 1-5 & 8-12
- Arm C: Relapsed AML, MDS and MF: AZD1775 only
  Relapsed/Refractory AML & HMA failure AML/ MDS and Relapsed/Refractory Primary & Secondary MF
  AZD1775 only: AZD1775 days 1-5 & 8-12
Period: Overall Study
Arm/Group | Arm A: Elderly Newly Diagnosed AML | Arm B:Relapsed AML and MDS | Arm C: Relapsed AML, MDS and MF
Started | 3 | 2 | 1
Completed | 0 | 0 | 0
Not Completed | 3 | 2 | 1
Not completed — Death | 1 | 0 | 0
Not completed — Progression of Disease | 1 | 0 | 0
Not completed — Withdrawal of Informed Consent | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total Participants: Participants from all 3 arms:
  Arm A: Elderly Newly Diagnosed AML Arm B: Relapsed AML and MDS Arm C: Relapsed AML, MDS, and MF
  Baseline information cannot be separated by diagnoses due to data privacy reasons
Arm/Group | Total Participants
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 2
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission (CR) Rate
Description: Less than 5% blasts in a non-hypocellular marrow with a granulocyte count ≥ 1.0, and a platelets count of ≥ 100 with complete resolution of extramedullary disease and absence of peripheral blood blasts.
Time Frame: 4 months
Population: No data was collected for this outcome measure due to early termination of study.
Arm/Group | Arm A: Elderly Newly Diagnosed AML | Arm B:Relapsed AML and MDS | Arm C: Relapsed AML, MDS and MF
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Incomplete Measure of Complete Remission (CRi)
Description: is called if patient meets all CR criteria except for residual neutropenia (ANC<1 x109/L) or thrombocytopenia (platelets<100 x109/L)
Time Frame: 4 months
Population: No data was collected for this outcome measure due to early termination of study.
Arm/Group | Arm A: Elderly Newly Diagnosed AML | Arm B:Relapsed AML and MDS | Arm C: Relapsed AML, MDS and MF
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Complete Cytogenetic Remission (CCyR)
Description: The absence of chromosome abnormalities (if present at diagnosis) on conventional cytogenetic study using G-banding (at least 10 metaphases present).
Time Frame: 4 Months
Population: No data was collected for this outcome measure due to early termination of study.
Arm/Group | Arm A: Elderly Newly Diagnosed AML | Arm B:Relapsed AML and MDS | Arm C: Relapsed AML, MDS and MF
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Arm A: Elderly Newly Diagnosed AML | Arm B:Relapsed AML and MDS | Arm C: Relapsed AML, MDS and MF
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Elderly Newly Diagnosed AML (N=3) | Arm B:Relapsed AML and MDS (N=2) | Arm C: Relapsed AML, MDS and MF (N=1)
Progression of Disease (General disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-23): https://cdn.clinicaltrials.gov/large-docs/43/NCT03718143/Prot_SAP_000.pdf